CLINICAL TRIAL: NCT00427024
Title: Study of Renal Transporters and Their Regulators After Renal Transplantation
Brief Title: Renal Transporters After Renal Transplantation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Muenster (Other)
Other Study IDs: NTX + Transport
Record Dates: First submitted 2007-01-25; First posted 2007-01-26 (Estimated); Last update posted 2007-02-06 (Estimated); Status verified 2007-02

CONDITIONS: Kidney Transplantation; Host vs Graft Reaction
Keywords: renal transplantation; acute rejection; transport; transporter; acute rejection after renal transplantation

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Previous studies in animals revealed, that the activity of certain transporters along the nephron is changed with acute rejection after renal transplantation. We intend to investigate underlying mechanisms occurring in man in renal biopsy specimens obtained from patients because of acute rejection of the transplant or chronic transplant nephropathy.

DETAILED DESCRIPTION:
After renal transplantation, caused by ischemia or rejection, often renal transport processes are disturbed. These dysfunctions which are similar to the Fanconi syndrome as well as renal tubular acidosis occur in the early phase after transplantation. Irreversible injuries develop caused by nephrotoxicity of immunosuppressants and renal transplant artery stenoses. Although this has impact on clinical follow up and prognosis of the transplant, up to now, it still has to be clarified by which mechanisms the tubular transport processes are impaired.

In an animal model, we demonstrated first, that expression of membrane proteins is specifically modulated early after transplantation, indicating that changes in expression and function in these models are not due to general necrosis or apoptosis. Second, our results differ from data obtained after ischemia / reperfusion. Third, the regulatory pattern seems not to be the consequence of a systemic effect. We suppose that changes in expression of transporters and receptors after transplantation and rejection are continuously modulated, which may influence the prognosis of the graft. The data suggest that transplantation with acute rejection leads to ischemia-independent changes in the regulation of transporters along the nephron (Velic A, Gabriëls G, Hirsch JR, Schröter R, Edemir B, Paasche S, Schlatter E. Acute rejection after rat renal transplantation leads to downregulation of Na+ and water channels in the collecting duct. Am J Transplant. 2005, 5: 1276-85. Velic A, Hirsch JR, Bartel J, Thomas R, Schröter R, Stegemann H, Edemir B, August C, Schlatter E, Gabriëls G: Renal transplantation modulates expression and function of receptors and transporters of rat proximal tubules. J Am Soc Nephrol. 2004, 15: 967-77).

By means of microarray analysis we examined the expression of genes after renal transplantation in rats. Of the about 18.000 genes, in the model of acute rejection more than 55% of the genes were changed in their expression compared to controls, while transplantation without rejection only induced a change in expression of 30% of the genes. With rejection, about 50% of these genes were upregulated and about 50 % downregulated.

The regulated genes were classified in different groups. An essential part of the genes upregulated with rejection, as expected, point to a massive immune response. With rejection, a large amount of the genes coding for proteins with transport activity or proteins involved in metabolism are downregulated (e.g. amino acid transport, glucose transport, K+-, Ca++- and phosphate transport, transport of water, pH regulation). It was shown that, with rejection, signal transduction pathways involved in protein catabolism and immune response are upregulated.

By the present study in renal biopsies of about 200 transplanted individuals with acute rejection or chronic transplant nephropathy, we intend to examine the regulation of transport systems and regulatory factors during a period of two years. Our hypothesis is that the activity of transporters along the nephron is changed with renal transplantation, acute rejection reaction, or chronic transplant nephropathy. We intend to investigate underlying mechanisms in renal biopsy specimens obtained from patients because of acute rejection reaction or chronic transplant nephropathy.

The study has been designed to analyze whether the renal transport system factors we found to be differentially regulated in rats are regulated similarly with transplant rejection or transplant nephropathy in man.

The findings obtained by these studies also are indispensable regarding a plain comprehension of the development of tubule dysfunction after renal transplantation in man. The examination of the material serves to explore basic pathophysiological mechanisms with rejection and transplant nephropathy.

Details

Individuals with a renal transplant in whom a renal biopsy is indicated because of clinical reasons will be informed about aims and course of the study as well as potential risks and complications of the biopsy procedure. Then they will be asked to participate.

Should the patient decide for participation, he again will be made aware about potential risks and complications of the biopsy procedure using the official information sheet of the hospital on biopsy procedures and a special information sheet affiliated to the study documents. After reading the information sheets, the patients will be asked to sign the agreement. With the patients´ approval, two specimens of the renal transplant will be obtained. The Patient will be monitored for 24 hours clinically and by blood pressure measurements, urinalysis as well as by ultrasound scanning.

If there are no complaints and the controls are alright, the patient may check out of the hospital but is asked to return for a control examination one week later. At this presentation a physician familiar with the study will examine the patient clinically and by ultrasound. The levels of electrolytes, BUN and serum-creatinine will be detected and a venous blood gas analysis will be performed. In case that regarding the consequences of the biopsy everything is fine, the study is finished for this patient. He will be asked to present again, if new symptoms will arise.

While one part of the specimens obtained for diagnostics will be prepared for the study of gene expression immediately after the biopsy procedure, the other will be transported to the institute of pathology and worked up as usual.

ELIGIBILITY:
Inclusion Criteria:

* individuals transplanted with a donor kidney
* individuals with acute transplant rejection

Exclusion Criteria:

* pregnancy
* malignant disease
* HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2007-02; Study Completion 2009-02

CONTACTS AND LOCATIONS:
Overall Officials: Gert Gabriëls, PD Dr. med., Study Chair — University Hospital Münster
Locations (1):
- University Hospital Münster, Münster, Germany

REFERENCES:
- [Background] Velic A, Gabriels G, Hirsch JR, Schroter R, Edemir B, Paasche S, Schlatter E. Acute rejection after rat renal transplantation leads to downregulation of NA+ and water channels in the collecting duct. Am J Transplant. 2005 Jun;5(6):1276-85. doi: 10.1111/j.1600-6143.2005.00890.x. PMID 15888031
- [Background] Velic A, Hirsch JR, Bartel J, Thomas R, Schroter R, Stegemann H, Edemir B, August C, Schlatter E, Gabriels G. Renal transplantation modulates expression and function of receptors and transporters of rat proximal tubules. J Am Soc Nephrol. 2004 Apr;15(4):967-77. doi: 10.1097/01.asn.0000117287.74203.89. PMID 15034099